CLINICAL TRIAL: NCT06570616
Title: Strategies for Controlling Unintentional Leakage in the Treatment of Obstructive Sleep Apnea With Continuous Positive Airway Pressure
Brief Title: Addressing Unintentional Leakage When Using Nasal CPAP - Study A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Pedro Rodrigues Genta, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: avniocpapn1
Record Dates: First submitted 2024-01-25; First posted 2024-08-26 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Continuous Positive Airway Pressure; Adverse Effect; Obstructive Sleep Apnea
Keywords: CPAP; Excessive leak; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant
Masking Description: CPAP device screen is taped to hide CPAP level and mode
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AutoCPAP (Experimental): Subjects will use auto CPAP during 7 days.
  Interventions: Device: APAP (automatic mode)
- Fixed (Experimental): Subjects will start with the CPAP level obtained during auto-CPAP titration. CPAP will be decreased according to the study protocol.
  Interventions: Device: CPAP (fixed mode)

INTERVENTIONS:
Device: CPAP (fixed mode) — Patients will undergo strategies to control excessive leakage while using autoCPAP vs. progressively decreasing fixed nasal CPAP. Before randomization, subjects will undergo an autoCPAP titration for 3 days. Subjects will then be randomized to start the protocol with autoCPAP or fixed CPAP and then will switch to the alternative arm.
  Arms: Fixed
Device: APAP (automatic mode) — Patients will undergo strategies to control excessive leakage while using autoCPAP vs. progressively decreasing fixed nasal CPAP. Before randomization, subjects will undergo an autoCPAP titration for 3 days. Subjects will then be randomized to start the protocol with autoCPAP or fixed CPAP and then will switch to the alternative arm.
  Arms: AutoCPAP

SUMMARY:
Oral unintentional leak is a common side effect of continuous positive airway pressure (CPAP) for obstructive sleep apnea (OSA) treatment. Management of oral unintentional leakage has not been standardized and the effectiveness of potential approaches have not been studied in controlled studies. Higher levels of CPAP are associated with higher leak. In the present study, a sequential approach to control excessive unintentional leak will be tested. In study A, the reduction of therapeutic CPAP level will be tested. In study B, oronasal CPAP will be compared to nasal CPAP with a chinstrap.

DETAILED DESCRIPTION:
Study A will consist of a cross-over controlled randomized trial to compare unintentional leak during auto-CPAP and during fixed CPAP after the progressive reduction of fixed CPAP, starting at the 90 th percentile obtained during a period of auto-CPAP. The order of interventions will be randomized. Auto-CPAP with a nasal mask will be used for 7 days. In the fixed CPAP arm, CPAP will be progressively reduced over a period of up to 21 days until leak is controlled or residual apnea-hypopnea index increases over 10 events/h. Subjects that persisted with excessive leak at the end of the Study A will be invited to Study B.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate and severe obstructive sleep apnea;
* Use of CPAP with a nasal mask;
* 95th percentile of unintentional leak from the last 7 days above 24 l/min or at least 4 sudden leak line drop events

Exclusion Criteria:

* Patients who experience unintentional leakage from the mask/accessories.
* Diagnostic polysomnography examination with a predominance of central apnea;
* Patients with unstable heart disease, bedridden, neurodegenerative diseases, severe psychiatric disorders and COPD;
* Previous surgery for obstructive sleep apnea;
* Severe nasal obstruction (NOSE questionnaire score equal or greater then 55 points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
95th CPAP unintentional leak | 27 days
  The 95th unintentional leak percentile value will be compared during both interventions

SECONDARY OUTCOMES:
CPAP Side-effects questionnaire | 27 days
  This questionnaire addresses CPAP side-effects including those related to excessive air leak using a visual-analog scale.

OTHER OUTCOMES:
CPAP level | 27 days
  CPAP level will be compared during both interventions
Residual apnea-hypopnea index (AHI) | 27 days
  Residual AHI will be compared during both interventions
Functional Outcomes of Sleep Questionnaire (FOSQ 10) | 27 days
  The FOSQ 10 aims to assess the impacts of daytime sleepiness on daily activities. The FOSQ 10 consists of 10 questions comprising 5 items: General productivity, alertness, activity level, social outcomes, and intimate and sexual relationships. Each item generates a score from 1 to 4, and for items with more than one question, the average of the scores is calculated. The overall score is given by multiplying the average of the item scores by 5, obtaining a value from 5 to 20. The higher the score, the better the individual's functional status.
Pittsburgh questionnaire | 27 days
  The Pittsburgh questionnaire assessed sleep quality over the past month. The questionnaire consists of 19 self-reported questions and 5 questions related to the roommate/bed partner that are not included in the overall score. The 19 self-reported questions are divided into 7 components (respectively, subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime sleep dysfunction), and each component is scored on a scale of 0 to 3. The scores are then summed to form an overall scale of 0 to 21 points. The higher the score, the worse the sleep quality, and a PSQI greater than 5 indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Genta, Principal Investigator — Study Principal Investigator
Locations (2):
- Brazil (2):
  - Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil
  - InCor - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No